CLINICAL TRIAL: NCT04624334
Title: Electro-Entero-Graphy (EEnG) for Non-invasive Diagnosis of Motility Disorders of the Bowel
Brief Title: Non-invasive Assessment of Colonic Motility
Acronym: non-CoMoti
Status: Terminated | Type: Observational
Why Stopped: Money issues
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 110933
Record Dates: First submitted 2020-10-29; First posted 2020-11-10 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-04

CONDITIONS: Colon Disease; Functional Constipation; Electroenterography; Slow Transit; Hirschsprung Disease
MeSH Terms: conditions — Colonic Diseases; Hirschsprung Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Children with motility disorder
  Interventions: Other: Elektro-Entero-Graphy procedure; Other: EEnG Questionnaire; Other: Gold Standard Questionnaire
- Healthy children
  Interventions: Other: Elektro-Entero-Graphy procedure; Other: EEnG Questionnaire
- Adults with motility disorder
  Interventions: Other: Elektro-Entero-Graphy procedure; Other: EEnG Questionnaire; Other: Gold Standard Questionnaire
- Healthy adults
  Interventions: Other: Elektro-Entero-Graphy procedure; Other: EEnG Questionnaire

INTERVENTIONS:
Other: Elektro-Entero-Graphy procedure — Fasting, after which pre- and postprandial EEnG measurements are performed.
Other: EEnG Questionnaire — Filling out questionnaire about EEnG procedure.
Other: Gold Standard Questionnaire — Filling out questionnaire about Gold Standard diagnostic used to diagnose colonic motility disorder.
  Groups: Adults with motility disorder; Children with motility disorder

SUMMARY:
The current diagnostic process of colonic motility disorders often takes a long time and involves multiple invasive, painful and/or unnecessary diagnostic procedures. To improve this diagnostic process, the potential of Electro-Entero-Graphy (EEnG) is investigated.

During the EEnG procedure, several surface electrodes are positioned (under ultrasound guidance) on the abdomen so that electrical activity originating in the colon can be measured. Measurements will be performed after a period of fasting (when the colon is 'silent') and just after a meal (when the colon is moving) in both participants suffering from colonic motility disorders and healthy controls.

It is hypothesized that these measurements are an indication of colonic motility and can be used as a diagnostic tool for colonic motility disorders. It is also hypothesized that this EEnG procedure is not more burdensome than the Gold Standard procedures for diagnosing colonic motility disorders. This will be assessed using questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* All participants:
* Age ≤ 11 years for babies and children
* Age ≥ 18 years for adults.

Patients

* For babies/children:

  * suffering from surgically untreated HSCR as determined by a rectal biopsy, or
  * suspected of HSCR, for which a rectal biopsy is planned
* For adults: Suffering from a (suspected,) surgically untreated functional colonic motility disorder (such as slow-transit constipation, idiopathic/therapy resistant constipation of the colon), as diagnosed previously or will be diagnosed in the near future using the gold standard method.

Exclusion criteria:

* All participants:
* For adults: BMI > 27 kg/m2
* For babies/children: weight for length > 2.5 standard deviations of WHO Child Growth Standard
* Pregnancy
* Diabetes
* Any food intolerance
* Presence of an intestinal stoma
* Use of continuous tube feeding
* Healthy controls:
* The presence of any known gastro-intestinal conditions
* Use of laxatives in the past two years
* Participants with (suspected) motility disorder:
* (Part of) colon removed
* Inflammatory bowel disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All subjects fulfilling the in- and exclusion criteria will be included. Participants with (suspected) motility disorder will be recruited mainly in the Radboudumc and with the help from the Hirschsprung's patient association.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Power Percent Difference | During EEnG procedure
  Relative power change when comparing pre-prandial EEnG measurements to post-prandial measurements. Power will be calculated as the mean amplitude (mV^2/Hz) in a bandwidth of 2 cycles per minute around the dominant frequency related to colonic movements (between 2-10 cycles per minute).

SECONDARY OUTCOMES:
EEnG questionnaire score | Directly after EEnG procedure, which is a one time procedure the subjects in this study will undergo
  Burden score of EEnG procedure as assessed by a self created questionnaire (in collaboration with medical doctors, a psychologist and representatives of the patients association). A mean score of 0 indicates maximum burden, a mean score of 10 means no burden at all.
Gold Standard questionnaire score | Directly after EEnG procedure, which is a one time procedure the subjects in this study will undergo, or directly after the gold standard procedure, which some subjects will undergo in the near future at time of inclusion
  Total burden score of Gold Standard procedure used to diagnose motility disorder as assessed by a self created questionnaire (in collaboration with medical doctors, a psychologist and representatives of the patients association). A mean score of 0 indicates maximum burden, a mean score of 10 means no burden at all.

CONTACTS AND LOCATIONS:
Overall Officials: S.M.B.I. Botden, MD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available to other researchers on reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After publication of the results.
Access Criteria: Upon reasonable request via e-mail.